CLINICAL TRIAL: NCT03784833
Title: A Registry Study of Biomarkers in Heart Failure
Acronym: BIOMS-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Tianjin Medical University Second Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Beijing Luhe Hospital (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMS-HF
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Diseases
Keywords: heart failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Blood Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry study aims to discover the prognostic value of bio-markers in heart failure

DETAILED DESCRIPTION:
The purpose of this study is to investigate the prognostic value of biomarkers in Heart Failure.Patients with confirmed diagnosis of heart failure are enrolled.The primary outcome is all-cause mortality based on the death certificates. The secondary outcome is readmission for heart failure and all-cause mortality/readmission for heart failure according to the patients' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at the time of admission to the hospital
* With symptoms of new-onset or worsening heart failure
* Received or is eligible to receive a principal hospital discharge diagnosis of HF
* With signs and syndromes as follows: dyspnea at rest or with minimal exertion (dyspnea, orthopnea, or edema)；Rales, peripheral edema, ascites, or pulmonary vascular congestion on chest radiography.
* Patients who received packed red blood cells, whole blood, or platelets less than 10 days before the blood sample was taken;

Exclusion Criteria:

* Have objective evidence of cardiac dysfunction documented either by plasma concentrations of BNP and/or N-terminal pro-brain natriuretic peptide (NT-proBNP) <35 pg/mL or <125 pg/ml, respectively
* Current known inability to follow instructions or comply with follow-up procedures.
* Eligible patients without informed consent form

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure accorrding to Inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Number of death (all cause) | 2 years of follow-up
  Number of death within 2 years of discharge

SECONDARY OUTCOMES:
Number of rehospitalizations for acute heart failure (HF) | 2 years of follow-up
  Number of heart failure related hospitalization within 2 years of discharge
Number of death ( all cause) or readmission for heart failure | 2 years of follow-up
  Number of Death or heart failure related hospitalization within 2 years of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, Dr, Study Director — The Key Laboratory of Remodeling-Related Cardiovascular Disease, Ministry of Education, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart,Lung and Blood Vessel Diseases
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China